CLINICAL TRIAL: NCT00874120
Title: Randomized, Placebo-Controlled, Double-Blind, Two-Way Crossover Study to Evaluate the Effects of Phenylephrine HCl Extended-Release Tablets 30 mg Compared to Placebo on Ambulatory Blood Pressure
Brief Title: Safety Study Comparing Phenylephrine HCL Extended Release Tablets 30 mg and Placebo (Study CL2007-07)(P07529)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 18121; CL2007-07; P07529 (Other: Merck)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Blood Pressure; Human Experimentation
MeSH Terms: interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine HCl Extended-Release tablets 30 mg (Experimental): Phenylephrine HCl Extended Release tablets 30 mg
  Interventions: Drug: Phenylephrine Hydrochloride (HCl) Extended-Release tablets 30 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenylephrine Hydrochloride (HCl) Extended-Release tablets 30 mg — Phenylephrine HCl Extended-Release tablets 30 mg taken twice daily (12 hours apart) for 7 days.
  Arms: Phenylephrine HCl Extended-Release tablets 30 mg
Drug: Placebo — Placebo taken twice daily (12 hours apart) for 7 days.
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled double-blind, crossover design study; 116 subjects randomized on Day 1 to obtain 98 completed subjects. Study will be composed of a 7-day period of therapy with randomized active or placebo treatment with a subsequent 6-8 day washout period, followed by a second 7-day period of double-blind therapy with the other agent. Ambulatory blood pressure measurement will be performed beginning on Day 7 of each treatment period following administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female volunteers must be 18 years or older, with a Body Mass Index (BMI) between 19-30 inclusive [BMI = weight (kilograms)/height (meters squared)].
* Clinical laboratory tests (complete blood count, blood chemistries, urinalysis), Human Immunodeficiency Virus (HIV) antibodies, hepatitis B surface antigen, hepatitis C antibody must be within normal limits or clinically acceptable to the Investigator/Sponsor.
* Drug screen for drugs and alcohol with a high potential for abuse must be negative at screening.
* Subjects must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations, procedures or participation.
* Subjects must agree not to take a monoamine oxidase inhibitor (MAOI) for two weeks (14 days) prior to study participation and for two weeks (14 days) after the end of their study participation.
* Subjects must have normal or clinically acceptable physical exam and Electrocardiogram (ECG) intervals (PR, QRS, QT and QTc) on 12-lead ECG (recorded at 25 millimeters/second [mm/s]).
* Subjects must have a mean after 5 minute of rest sitting systolic/diastolic office blood pressure ≤ 138/88 millimeters of mercury (mmHg).
* Subjects with controlled diabetes prior to entry must have a mean sitting after 5 minute of rest systolic/diastolic office blood pressure ≤ 128/78 mmHg from non-dominated arm
* Females must have the urine or serum pregnancy test (Human Chorionic Gonadotropin) that is negative at Screening and Day 1 of Period 1.
* Female subjects of childbearing potential must be using medically acceptable birth control measures.
* Subjects must understand the dosing schedule.
* Subjects must be able to read and write in English.

Exclusion Criteria:

* Subjects must not have any significant medical condition which, in the judgment of the Investigator, is a contraindication to the use of phenylephrine HCl, might interfere with the study or requires treatment expected to affect the blood pressure. These may include hyperthyroidism, hypothyroidism, uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease, elevated intraocular pressure, prostatic hypertrophy.
* Subjects who have a history of any clinically significant local or systemic infectious disease within four weeks prior to initial treatment administration.
* Subjects who have received an investigational drug within 30 days prior to study dosing.
* Subjects who are, appear to be, or are known, current or former drug addicts or alcoholics.
* Subjects who are positive for hepatitis B surface antigen or hepatitis C antibody.
* Subjects who are positive for HIV antibodies.
* Subjects who have a clinically significant history of food or drug allergy.
* Subjects who have a known allergy or intolerance to phenylephrine HCl.
* Females who are pregnant, nursing or unwilling to use/practice adequate contraception (hormonal, Intrauterine Device, barrier method, etc.).
* Subjects taking topical or oral decongestant products within 7 days of Visit 2.
* Subjects taking antihypertensive medication.
* Subjects taking monoamine oxidase inhibitors.
* Subjects taking tricyclic antidepressants (e.g. amitriptyline, nortriptyline, imipramine)
* Subjects taking antithyroid medication (e.g. propylthiouracil, methimazole, iodides).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenylephrine Followed by Placebo: Phenylephrine hydrochloride (HCl) Extended Release tablets 30 mg twice daily for 7 days followed by a 6- to 8-day washout period followed by placebo twice daily for 7 days
- Placebo Followed by Phenylephrine: Placebo twice daily for 7 days followed by a 6- to 8-day washout period followed by Phenylephrine HCl Extended Release tablets 30 mg twice daily for 7 days
Period: First Intervention
Arm/Group | Phenylephrine Followed by Placebo | Placebo Followed by Phenylephrine
Started | 58 | 58
Completed | 52 | 56
Not Completed | 6 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — positive drug test | 1 | 0
Period: Wash-out Period
Arm/Group | Phenylephrine Followed by Placebo | Placebo Followed by Phenylephrine
Started | 52 | 56
Completed | 52 | 56
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Phenylephrine Followed by Placebo | Placebo Followed by Phenylephrine
Started | 52 | 56
Completed | 50 | 56
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine Followed by Placebo | Placebo Followed by Phenylephrine | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.14) | 29.0 (10.99) | 29.2 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Average Systolic Blood Pressure (SBP) Readings for a 5-hour Range Around the Time of Maximum Concentration (Tmax).
Description: Five hour (hr) range around the Tmax was defined as approximately 2 hours before to approximately 2 hours after the Tmax, including Tmax. The parameters will be compared between active drug and placebo using analysis of variance (ANOVA). The 95% 2-sided Confidence Interval (CI) on the difference between treatments will also be presented.
Time Frame: 24 hours after final dose of each 7-day treatment period.
Population: The per-protocol population included 100 participants who completed both treatment periods and have 24-hour Ambulatory Blood Pressure Monitoring (ABPM) data for SBP measurements for each study drug, 46 participants who received phenylephrine followed by placebo and 54 participants who received placebo followed by phenylephrine.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Phenylephrine: Phenylephrine HCl Extended Release tablets 30 mg twice daily for 7 days
- Placebo: Placebo twice daily for 7 days
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 100 | 100
mmHg | 118.3 (9.24) | 118.6 (9.38)
Statistical Analysis 1: Comparison: Phenylephrine vs Placebo; Test type: Superiority or Other; p = 0.5480, ANOVA — P-value is based on an ANOVA model including sequence, subject within sequence, period and treatment as factors; residual error term from the ANOVA = -0.5, 95% CI 2-sided [-2.0 to 1.1]

ADVERSE EVENTS:
Description: Intent-to-treat population. Participants who received at least one dose of study medication were included in the safety population.
Arm/Group | Phenylephrine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/111
Other Adverse Events (participants affected / at risk) | 0/114 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves all publication and presentation rights.